ClinicalTrials.gov identifier: NCT02545114

Tolvaptan for patients with acute neurological injuries.

Main investigators: Kees H. Polderman, MD, PhD, and Brian T. Jankowitz, MD.

August 24<sup>TH</sup> 2018.

Study results

admission diagnosis of subarachnoid hemorrhage, one had an intracranial hemorrhage. The average dose of tolvapan given was 29.4mg. Sodium levels were 130.2±1.7 before tolvaptan, 132.3±3.4 at 12hrs, 135.4±3.1 at 24hrs, 137.2±3.5 at 48hrs, 136.1±3.4 at 72hrs, 137.8±2.9 at 96hrs, and 137.4±3.9 at 120hrs; the median treatment duration was 9 days. Enrollment was

Seventy-nine patients were screened, of whom 25 were enrolled; 24 of these patients had an

discontinued when 2 patients developed polyuria, persisting after tolvaptan discontinuation and likely unrelated to the drug; however, we deemed our screening process insufficient in excluding

CSW (the likely cause of polyuria) and decided to halt the current study and develop a new

protocol with better screening for CSW. No other adverse events occurred.